CLINICAL TRIAL: NCT02551068
Title: High Oxygen Delivery to Preserve Exercise Capacity in IPF Patients Treated With Nintedanib: The HOPE-IPF Study
Brief Title: High Oxygen Delivery to Preserve Exercise Capacity in Idiopathic Pulmonary Fibrosis Patients Treated With Nintedanib
Acronym: HOPE-IPF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Chrisopher Ryerson, MD, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H15-01200
Record Dates: First submitted 2015-09-01; First posted 2015-09-16 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Oxygen; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 60% Oxgyen (Experimental): While participants are exercising, they will be breathing 60% oxygen through a mask.
  Interventions: Other: 60% Oxygen
- Standard of Care (Placebo Comparator): While participants are exercising, they will be breathing air through a mask that will be titrated to keep oxygen saturation at least 88%, allowing a maximum inhaled oxygen percentage of 40%.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: 60% Oxygen — While participants are exercising, they will be inhaling 60% oxygen through a mask
  Arms: 60% Oxgyen
Other: Standard of Care — While participants are exercising, they will be breathing air through a mask that will be titrated to keep oxygen saturation at least 88%, allowing a maximum inhaled oxygen percentage of 40%.
  Arms: Standard of Care

SUMMARY:
The purpose is to determine if patients with idiopathic pulmonary fibrosis (IPF) taking nintedanib will have improved exercise endurance, breathlessness and quality of life if breathing 60% oxygen compared to standard of care during an 8 week exercise training program.

DETAILED DESCRIPTION:
Pulmonary rehabilitation is a structured evidence-based exercise and education intervention that is recommended for most patients with IPF. Pulmonary rehabilitation improves functional capacity (6-minute walk distance [6MWD]), breathlessness and quality of life in patients, however these benefits are often modest and only temporary. Nintedanib is an antifibrotic medication that has been shown to slow the decline of lung function. Use of antifibrotic medications in the pulmonary rehabilitation setting may therefore allow prolonged benefit of exercise training by preventing IPF progression and the resulting worsening symptoms and functional decline. Unpublished data suggest that breathing 60% oxygen in a pulmonary rehabilitation setting could enable patients to train at higher exercise intensities and thus derive greater physiological adaptations and clinical benefits compared with traditional pulmonary rehabilitation.

This is a randomized, blinded study with two arms (standard of care or 60% oxygen). The decision to start or stop treatment with nintedanib will be made by the participants treating physician based on clinical findings. If the treating physician decides to discontinue nintedanib, the participant will be allowed to continue in the study.

The exercise training program is 8 weeks long, with visits 3 times a week. In addition to the exercise training there are 13 visits occurring before, during and after the 8 week exercise training program. At study visits, participants will be required to conduct a 6 minute walk test and complete a quality of life questionnaire. Select study visits will also require lung function tests and exercise tests to be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Idiopathic Pulmonary Fibrosis (IPF) diagnosis according to American Thoracic Society and/or European Respiratory Society consensus criteria
* Appropriate candidate for pulmonary rehabilitation
* prescribed nintedanib by their treating physician or currently on nintedanib
* 6 minute walk distance 50m or more
* Oxygen saturation 92% or more by pulse oximetry at rest while breathing room air
* Clinically stable for the preceding 6 weeks

Exclusion Criteria:

* Contraindication to treatment with nintedanib (based on Canadian labeling)
* Contraindication to exercise testing (e.g. significant cardiovascular, musculoskeletal, neurological disease)
* Other significant extra-pulmonary disease that, based on clinical assessment, could impair exercise capacity and/or oxygenation
* Forced vital capacity (FVC) less than 50% or Diffusion capacity for carbon monoxide (DLCO) less than 25%
* Concurrent or recent participation (less than 6 months) in a pulmonary rehabilitation program
* Use of prednisone greater than 10 mg/day for more than 2 weeks within 3 months of the first study visit
* Use of pirfenidone within 4 weeks of screening
* Significant emphysema (less than 10% volume on high resolution computed tomography (HRCT) or forced expiratory volume at one second (FEV1)/FVC less than 0.70)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2015-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in exercise duration during the constant load exercise test at 8 weeks | 8 weeks
  An constant load exercise test on a stationary bike will be performed. Patients will be told to exercise for as long as possible and endurance time will be defined as the duration of the constant load exercise test.

SECONDARY OUTCOMES:
Change in 6 Minute Walk Distance (6MWD) at 8 weeks | 8 weeks
  Patients will be asked to walk, at their own pace, as far as they can in 6 minutes.
Change in the amount a patient is troubled by their breathlessness at 8 weeks | 8 weeks
  Measured using the modified Medical Research Council dyspnea scale (mMRC)
Change in the amount a patient is troubled by their breathlessness during the 6 Minute Walk Distance test at 8 weeks | 8 weeks
  Measured using the 10-point Borg scale during 6MWD
Change in the amount a patient is troubled by their breathlessness during the cycle exercise test at 8 weeks | 8 weeks
  Measured using the 10-point Borg scale during cycle exercise tests
Change in how much shortness of breath the patient experiences while doing normal activities at 8 weeks | 8 weeks
  Measured using the University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ).
Change in the amount of physical work a patient can do before becoming breathless at 8 weeks | 8 weeks
  Measured using the oxygen cost diagram (OCD).
Patient reported change in amount of physical activity at 8 weeks | 8 weeks
  Physical activity will be measured using the long form of the international physical activity questionnaire (IPAQ-LF).
Change in amount of physical activity at 8 weeks | 8 weeks
  Physical activity will be measured objectively using the Fit Bit activity monitor.
Change in Quality of Life at 8 weeks | 8 weeks
  Disease-specific quality of life will be measured using the St. George's Respiratory Questionnaire (SGRQ).

CONTACTS AND LOCATIONS:
Overall Officials: Chris Ryerson, MD, Principal Investigator — St. Paul's Hospital; Jordan Guenette, PhD, Principal Investigator — St. Paul's Hospital
Locations (8):
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - UBC Okanagan, Kelowna, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Queens University, Kingston, Ontario
  - McGill University, Montreal, Quebec
  - Laval University, Québec

REFERENCES:
- [Derived] Ryerson CJ, Camp PG, Eves ND, Schaeffer M, Syed N, Dhillon S, Jensen D, Maltais F, O'Donnell DE, Raghavan N, Roman M, Stickland MK, Assayag D, Bourbeau J, Dion G, Fell CD, Hambly N, Johannson KA, Kalluri M, Khalil N, Kolb M, Manganas H, Moran-Mendoza O, Provencher S, Ramesh W, Rolf JD, Wilcox PG, Guenette JA. High Oxygen Delivery to Preserve Exercise Capacity in Patients with Idiopathic Pulmonary Fibrosis Treated with Nintedanib. Methodology of the HOPE-IPF Study. Ann Am Thorac Soc. 2016 Sep;13(9):1640-7. doi: 10.1513/AnnalsATS.201604-267OC. PMID 27348402